CLINICAL TRIAL: NCT04632589
Title: Angiotensin II Receptor Inhibition to Improve Microvascular Function in Women Who Have Had Preeclampsia
Brief Title: Losartan for Improved Vascular Endothelial Function After Preeclampsia
Acronym: LIVE-PE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anna Stanhewicz, PhD (Other)
Responsible Party: Sponsor-Investigator, Anna Stanhewicz, PhD, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 202006148
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Preeclampsia Postpartum
MeSH Terms: interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Losartan (Experimental): 6 weeks of daily (50mg/day) oral losartan potassium tablet
  Interventions: Drug: Losartan Potassium
- Placebo (Placebo Comparator): 6 weeks of daily oral placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan Potassium — subjects ingest 50mg losartan potassium tablet daily for 6 weeks
  Arms: Losartan
Drug: Placebo — subjects ingest placebo tablet daily for 6 weeks
  Arms: Placebo

SUMMARY:
Women who develop preeclampsia during pregnancy are more likely to develop and die of cardiovascular disease later in life, even if they are otherwise healthy. The reason why this occurs is unclear but may be related to blood vessel damage and increased inflammation that occurs during the preeclamptic pregnancy and persists postpartum. The purpose of this investigation is to determine the mechanisms contributing to this lasting blood vessel damage and to test whether taking a medication that blocks angiotensin II receptors (losartan) decrease these negative effects in women who have had preeclampsia. Identification of these mechanisms and treatment strategies may lead to better clinical management,of cardiovascular disease risk in these women.

In this study we use the blood vessels in the skin as a representative vascular bed. Using a minimally invasive technique (intradermal microdialysis for the local delivery of pharmaceutical agents) we examine the blood vessels in a nickle-sized area of the skin in women who have had preeclampsia. We make these measurements after the subjects take a placebo and after they take losartan (an angiotensin II receptor blocker) to test whether this treatment improves vascular function in these women. As a compliment to these measurements, we also draw blood from the subjects and isolate the inflammatory cells to test how sensitive their inflammatory responses are following the placebo and the losartan treatment.

ELIGIBILITY:
Inclusion Criteria:

Post-partum women,

* 18 years or older,
* who have delivered within 24 months of the study visit
* who have had a preeclamptic pregnancy diagnosed by their obstetrician and confirmed according to the American College of Obstetricians and Gynecologists criteria for preeclampsia. [This information will be self-reported by the subjects.]
* Using an effective method of birth control and not planning to become pregnant in the next 6 months.

Exclusion Criteria:

* skin diseases,
* current tobacco use,
* diagnosed or suspected hepatic or metabolic disease including chronic kidney disease (CKD) defined as reduced eGFR < 60 mL/min/1.73m2,
* statin or other cholesterol-lowering medication,
* current antihypertensive medication,
* history of hypertension prior to pregnancy,
* history of gestational diabetes,
* current pregnancy or breastfeeding,
* body mass index <18.5 kg/m2,
* allergy to materials used during the experiment.(e.g. latex),
* known allergies to study drugs.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2020-11-22 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Stanhewicz, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Losartan Than Placebo: 6 weeks of daily (50mg/day) oral losartan potassium tablet followed by 14 day washout period then 6 weeks of daily oral placebo tablet.
  Losartan Potassium: subjects ingest 50mg losartan potassium tablet daily for 6 weeks Placebo: subjects ingest placebo tablet daily for 6 weeks
- Placebo Than Losartan: 6 weeks of daily oral placebo tablet followed by 14 day washout period then 6 weeks of daily oral placebo tablet.
  Placebo: subjects ingest placebo tablet daily for 6 weeks Losartan Potassium: subjects ingest 50mg losartan potassium tablet daily for 6 weeks
Period: Overall Study
Arm/Group | Losartan Than Placebo | Placebo Than Losartan
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants were randomized to receive both interventions.
Arm/Group | All Study Participants
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Cutaneous Conductance (%Maximum) Response to Acetylcholine
Description: Cutaneous vascular vasodilator response to exogenous acetylcholine perfusion; measured with laser-Doppler flowmetry during intradermal microdialysis delivery of acetylcholine alone or co-infused with L-NAME. Cutaneous conductance is calculated (laser-Doppler flux/mean arterial pressure) and normalized to site specific maximal dilation (%maximum).
Time Frame: immediately following 6 weeks of oral treatment (losartan or placebo)
Population: All participants completed both treatments in randomized, blinded, cross-over design
Measure: Mean (Standard Deviation); unit: % of maximal cutaneous conductance
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 11 | 11
% of maximal cutaneous conductance | 89.4 (22.6) | 72.5 (16.5)

2. Primary Outcome: Cutaneous Conductance (%Baseline) Response to Angiotensin II
Description: Cutaneous vascular constrictor response to exogenous ang II perfusion; measured by laser-Doppler flowmetry during intradermal microdialysis delivery of angiotensin II. Cutaneous conductance is calculated (laser-Doppler flux/mean arterial pressure) and normalized to site-specific baseline conductance (%baseline) measured on the study day before the perfusion of angiotensin II.
Time Frame: immediately following 6 weeks of oral treatment (losartan or placebo)
Population: all participants completed both treatments in randomized, blinded, cross-over design
Measure: Mean (Standard Deviation); unit: % of baseline cutaneous conductance
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 11 | 11
% of baseline cutaneous conductance | 76.7 (29.1) | 53.8 (27.3)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected weekly (weeks 1, 2, 3, 4, 5, and 6) during each 6 week treatment period (placebo and losartan) for a total of 12 weeks. Adverse event data were not collected during the 2 week washout period between treatments.
Arm/Group | Losartan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT04632589/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT04632589/ICF_001.pdf